CLINICAL TRIAL: NCT06737783
Title: Effects of Thoracic Mobility Exercises on Thoracic Hyper Kyphosis and Impact on Hamstring Flexibility in Patients With Tibio Femoral Arthritis
Brief Title: Thoracic Mobility Exercises Impact in Tibio Femoral Arthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/02007 Sameen Fatima
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis (Knee OA)
Keywords: Thoracic hyperkyphosis; Hamstring flexibility; thoracic mobility exercises
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic mobility exercises + Conventional therapy (Experimental): mobility exercises comprises of Cat and camel stretch (On hands and knees (supported with knee braces), alternating between arching the back up and dropping it down to stretch thoracic spine), Thoracic rotations in side lying (side lying on the side with knees bent, rotating the upper body to increase thoracic mobility alternatively), Thoracic extension at wall using body weight (Standing with back to wall, gently pushing the upper back into extension while keeping the lower back stable), half kneeling chop thrust (Kneeling on one knee (supported with knee braces), rotating the torso while keeping the pelvis stable to mobilize the thoracic spine) ,Thoracic extension with a foam roller (Lying on the back with foam roller along thoracic spine, rolling gently to extend the thoracic spine in supine position). Adopt these positions with 5 secs hold and 15-20 reps will be performed for 2 sets and 10 reps per set.
  hold and 15-20 reps will be performed for 2 sets and 10 reps per set.
  Interventions: Other: Thoracic mobility exercises + Conventional therapy
- Self myofascial release with foam roller, T6- T7 Maitland mobilization and conventional therapy (Active Comparator): Hamstring Self myofascial release with foam roller (Sitting with one leg extended, roll the foam roller along the hamstring while applying pressure to tender spots) 3 sets with 30 to 120 secs rolling duration per second for 5 mins T6-T7 grade 3 Maitland mobilization (Lying on the back, the therapist applies a sustained, posterior-to-anterior force on T6-T7 in prone position) 30 repetitions, with 1 min rest between 4 sets for 15 mins.
  Conventional therapy includes Hot pack/Cold pack + tens = 15 mins, Frequency 80 Hz, Pulse duration: 100 microseconds, Static quads (10 reps, 10 second hold, 2 sets), Active knee flexion and extension ROMs (10 reps, 5 secs hold, 2 sets), Long Axis Knee traction (5 reps, 30 secs hold, 10sec rest in b/w 2 sets), Kaltenborn Knee Glides Ant and Post direction ( 5 reps, 30 secs hold,10 sec rest interval in b/w 2 sets), Calf stretches (10 reps, 5 secs hold , 2 sets).
  Interventions: Other: Self myofascial release with foam roller, T6- T7 Maitland mobilization + Conventional therapy

INTERVENTIONS:
Other: Thoracic mobility exercises + Conventional therapy — mobility exercises comprises of Cat and camel stretch (On hands and knees (supported with knee braces), alternating between arching the back up and dropping it down to stretch thoracic spine), Thoracic rotations in side lying (side lying on the side with knees bent, rotating the upper body to increase thoracic mobility alternatively), Thoracic extension at wall using body weight (Standing with back to wall, gently pushing the upper back into extension while keeping the lower back stable), half kneeling chop thrust (Kneeling on one knee (supported with knee braces), rotating the torso while keeping the pelvis stable to mobilize the thoracic spine) , Thoracic extension with a foam roller (Lying on the back with foam roller along thoracic spine, rolling gently to extend the thoracic spine in supine position). Adopt these positions with 5 secs hold and 15-20 reps will be performed for 2 sets and 10 reps per set.
  Arms: Thoracic mobility exercises + Conventional therapy
Other: Self myofascial release with foam roller, T6- T7 Maitland mobilization + Conventional therapy — Hamstring Self myofascial release with foam roller (Sitting with one leg extended, roll the foam roller along the hamstring while applying pressure to tender spots) 3 sets with 30 to 120 secs rolling duration per second for 5 mins T6-T7 grade 3 Maitland mobilization (Lying on the back, the therapist applies a sustained, posterior-to-anterior force on T6-T7 in prone position) 30 repetitions, with 1 min rest between 4 sets for 15 mins. Conventional therapy includes Hot pack/Cold pack + tens = 15 mins, Frequency 80 Hz, Pulse duration: 100 microseconds, Static quads (10 reps, 10 second hold, 2 sets), Active knee flexion and extension ROMs (10 reps, 5 secs hold, 2 sets), Long Axis Knee traction (5 reps, 30 secs hold, 10sec rest in b/w 2 sets), Kaltenborn Knee Glides Ant and Post direction ( 5 reps, 30 secs hold,10 sec rest interval in b/w 2 sets), Calf stretches (10 reps, 5 secs hold , 2 sets).
  Arms: Self myofascial release with foam roller, T6- T7 Maitland mobilization and conventional therapy

SUMMARY:
The aim of this randomized clinical trial is to find the effect of thoracic mobility exercises on thoracic hyper kyphosis and hamstring flexibility with tibiofemoral arthritis patients on reducing hyper kyphotic posture, knee pain and improving flexibility of hamstring muscles.

DETAILED DESCRIPTION:
Tibio Femoral Arthritis is a painful heterogeneous musculoskeletal condition that comprises of articular cartilage degradation, distortion of joint tissues, depletion in synovial fluid and progression over time. Decline in joint ROM usually began in fourth decade, more common in women in the age of menopause mostly the age of 45 years or elder. In Pakistan prevalence of Tibio femoral arthritis is 28.0% in urban population and 25.0% in the rural population, estimated o outstretch 35% by 2030. Hamstring muscle are part of superficial posterior anatomical chain in body that form meridians or myofascial chains connected to thoracolumbar fascia via sacro tuberous ligament.

Knee joint movements are primarily facilitated by the quadriceps and hamstrings, which play a crucial role in ensuring smooth and accurate ambulation. Tightness in hamstring put stress on Tibio-femoral joint which further reduce its range of motion especially knee extension, joint loading problems, induce compensatory movements, gait limitations, disturbs overall spinal postural alignment, increase thoracic kyphosis, decrease lumbar lordosis, and inducing posterior pelvic tilt. Until now most existing studies focus on the impact of thoracic mobility on thoracic spine issues or general posture, with limited research on its secondary effects on lower limb flexibility in 45 to 65 years old Tibio femoral arthritic patients. There is still research gap present to identify comprehensive effects of thoracic mobility exercises, on hyper kyphotic postures with tightened hamstrings, complementing Tibio femoral arthritis with aging.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic Kyphotic angle > 40
* Asymptomatic (no pain symptoms in) thoracic spine
* Able to stand independently
* Less than 70 degree Hip Flexion Angle on active SLR, with limited knee extension range more than 20 degree restriction on AKE test
* Bilateral Hamstring tightness
* Visual Analogue Scale in targeted Joint Tibiofemoral arthritis >3 cm
* Having Osteoarthritis in Tibio femoral Joint, according to KL (Grade 2 and 3)
* X-rays showing evidence of reduced knee spaced/osteoarthritis symptoms B/L( >2 year)

Exclusion Criteria:

* Muscle/tendon injuries of hamstring
* Spinal Injuries, scoliosis, tumors and malignancies
* Any surgery, infection, skin sensitivity, trauma, fracture and fall
* Involvement in regular flexibility yoga program
* Patient with intra articular steroidal therapy with in last 6 months
* Patient unwilling to comply follow up schedule
* Patient involvement in another interventional study

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Active knee extension test (Goniometer) | 4 weeks
  Active knee extension (AKE) test was to measure hamstring flexibility. The participants lay in the supine/prone position with the tested hip flexed 90°, knee flexed 90° and were asked to extend the knee as much as possible until they felt strong resistance. Ensure Lumbar spine should be in neutral position. Axis of Goniometer will be placed on Lateral femoral condyle of femur. While moving and stationary arm on lateral aspect of midline of femur and fibula. Complete knee extension was 0° shows optimal flexibility and any lack of knee extension was measured with a universal goniometer with higher angle 20 degrees indicates poorer flexibility of hamstring muscles.
Visual Analogue scale VAS | 4 weeks
  The VAS is a simple bidirectional graphic tool with a 10-cm horizontal line for assessing musculoskeletal pain intensity. Left side of scale represent 0 digit indicates "no pain" and the right end marked with 10 indicates "worst imaginable pain". The participants were asked to draw a vertical mark on the line to represent their level of pain intensity when patient asked to extend knee from flexion and from flexion position to extension. The length from the left end to the vertical mark, made by the participant shown her/his pain intensity
Baseline bubble Inclinometer | 4 weeks
  Thoracic kyphosis angle was calculated using a baseline bubble inclinometer, a device used to measure curvature of spine. Inclinometer can measure angles b/w 20 to 60 degrees for thoracic region on wider arc of 180 degree. Participant should be in neutral position. Firstly, an inclinometer was placed over the spinous process of T1 and T2 for measurement (first inclinometer angle). Secondly, another inclinometer was placed over the spinous process of T12 and L1 for angle measurement (second inclinometer angle). The kyphosis angle was taken by taking difference between two measurements. Threshold for hyperkyphotic is greater 40 degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Maria khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- National Institue of Rehabilitation Medicine (Nirm), Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No